CLINICAL TRIAL: NCT02779946
Title: Non-invasive Liver Screening for Risk Assessment for Coronary Heart Disease
Acronym: NILS-R-CHD
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Universitätsklinikum Leipzig (Other)
Responsible Party: Principal Investigator, Sebastian Beer, Specialist in Internal Medicine, Principle Investigator, University of Leipzig
Other Study IDs: AD2-0401; 01EO1501 (Other Grant/Funding Number: Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2015-10-16; First posted 2016-05-23 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Coronary Disease; Non-alcoholic Fatty Liver Disease; Elasticity Imaging Techniques
MeSH Terms: conditions — Coronary Disease; Non-alcoholic Fatty Liver Disease | interventions — adiponutrin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CHD-positive: positive tested for coronary artery disease
  Interventions: Device: Fibro Scan; Genetic: PNPLA3
- CHD-negative: negative tested for coronary artery disease
  Interventions: Device: Fibro Scan; Genetic: PNPLA3

INTERVENTIONS:
Device: Fibro Scan
Genetic: PNPLA3

SUMMARY:
Background: Non-alcoholic fatty liver disease (NAFLD) is the hepatic manifestation of the metabolic syndrome, which is one of the major risk factors of coronary heart disease (CHD). CHD is the most important manifestation of atherosclerosis, because of its immense morbidity and mortality. Transient elastography (TE, Fibroscan®) including the currently developed controlled attenuation parameter (CAP) is a non-invasive method for evaluation of liver fibrosis and steatosis, which is already implemented in routine care of patients with NAFLD. Hypothesis: The use of TE with CAP as screening for NAFLD might be an easy tool for risk assessment for CHD. Methods: Patients scheduled for routine coronary angiography will be screened for manifestation of NAFLD by TE including CAP, conventional ultrasound, clinical and laboratory parameters. Patients will be stratified for the presence of CHD based on the angiography results and correlation analysis with liver fat content will be performed. NFALD screening will be validated in a subgroup by MR-based measurements.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age ≥ 18 years
* patients with indication for routine coronary angiography

Exclusion Criteria:

* transplanted liver
* resection of right liver lobe
* transaminases of > 5-fold upper limit
* pregnancy or lactation
* choleastasis on ultrasound imaging
* active malignant or consuming disease 12 month before inclusion
* congestive heart failure (EF<30%, NYHA III or IV, diastolic dysfunction °III or IV
* pulmonary hypertension (WHO °III or IV) Exclusion criteria for MR diagnostics
* pacemaker or ICD
* non removable magnetizable metal implants
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for routine angiography of coronary vessles to the Division of cardiology and angiography of the University Hospital Leipzig
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Correlation of presence CHD and NAFLD | 1 year
  Routine angiography defines the presents of CHD. Fibroscan will determine whether and to which extent a NAFLD is present.

SECONDARY OUTCOMES:
Correlation of severity of CHD and NAFLD | 1 year
  Correlation of severity of CHD defined by angiography (Multi or Single vessel disease) will be correlated by quantification of liver fibrosis and steatosis on Fibroscan.
Fibrocan vs MR-based methods | 1 year
  MRS will be evaluated and correlated to the results of Fibroscan in a subset of patients.
Correlation of NAFLD and intima media thickness | 1 year
  intima media thickness of the common carotid artery is correlated to the Fibroscan results
Correlation of NAFLD and other signs of atherosclerosis | 1 year
  Plaque burden of abdominal aorta and carotid artery will be correlated to the results of Fibroscan.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Beer, MD, Principal Investigator — Leipzig University Medical Center, IFB AdiposityDiseases
Locations (1):
- Leipzig University Medical Center, Leipzig, Germany